CLINICAL TRIAL: NCT01068080
Title: Prediction of Impaired Myocardial Fatty Acid Metabolism and Insulin Resistance for Cardiac Death of Hemodialysis Patients With Normal Coronary Arteries
Brief Title: Involvement of FFA Metabolism and Insulin Resistance in Cardiac Death
Acronym: CD_HD_FAIR
Status: Completed | Type: Observational
Sponsor: Toujinkai Hospital (Other)
Responsible Party: Masato Nishimura, MD, PhD, Toujinkai Hospital
Other Study IDs: Toujinkai Clincal Study-2
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2000-10

CONDITIONS: Kidney Disease; Coronary Artery Disease; Hemodialysis
Keywords: fatty acid metabolism; insulin resistance; cardiac death; hemodialysis; normal coronary arteries; Predictive values of impaired myocardial fatty acid metabolism or insulin resistance for cardiac death of hemodialysis patients with normal coronary arteries
MeSH Terms: conditions — Kidney Diseases; Coronary Artery Disease; Insulin Resistance; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myocardial fatty acid metabolism, Insulin resistance: Myocardial fatty acid metabolism was evaluated by myocardial fatty acid imaging using BMIPP SPECT.
  Insulin resistance was evaluated by HOMA-IR.

SUMMARY:
The investigators evaluated predictive values of myocardial fatty acid metabolism and insulin resistance for cardiac death of hemodialysis patients with normal coronary arteries.

DETAILED DESCRIPTION:
Dialysis patients have extraordinarily high mortality rates. Cardiac diseases play an important role in deaths among end-stage renal disease (ESRD) patients undergoing renal replacement therapy. Previous studies have shown that maintenance hemodialysis patients have high prevalence of obstructive coronary artery disease. While obstructive coronary artery disease is undoubtedly involved in cardiac deaths induced by acute myocardial infarction or congestive heart failure and in sudden cardiac death, cardiac death can occur in hemodialysis patients who have apparently no pre-existing obstructive coronary artery disease. However, few studies have investigated the factors which are useful for stratifying the risk of cardiac death in dialysis patients with normal coronary arteries.

We recently showed that visualizing severely impaired myocardial fatty acid metabolism on images can help not only to detect obstructive coronary artery disease [8], but also to identify patients at high risk of cardiac death among hemodialysis patients without coronary intervention or old myocardial infarction and among those with coronary revascularization by percutaneous coronary artery intervention. In addition, combination of impaired cardiac fatty acid metabolism with insulin resistance, which is one of the risk factors related with coronary atherosclerosis, may contribute to left ventricular dysfunction in patients with maintenance hemodialysis with normal coronary arteries. Impaired myocardial fatty acid metabolism and insulin resistance, both of which reduce the synthesis of myocardial adenosine triphosphate (ATP), are likely to be involved in fatal cardiac events by causing deficiency of myocardial energy supply. In this study, we prospectively investigated the potential of myocardial fatty acid metabolism and insulin resistance to predict cardiac death in hemodialysis patients without pre-existing obstructive coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients who had normal coronary arteries identified by coronary angiography and underwent the examination of BMIPP SPECT and measurement of HOMA-IR as a parameter of insulin resistance.

Exclusion Criteria:

* Patients who had not done BMIPP SPECT within one month of coronary angiography
* Congestive heart failure (NYHA 3-4)
* Significant valvular heart disease
* Pacemaker
* Idiopathic cardiomyopathy
* Malignancy
* Patients who had not measured HOMA-IR within one month after coronary angiography
* Patients receiving extrinsic insulin or medication of sulfonylurea

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients who had normal coronary arteries identified by coronary angiography and underwent the examination of BMIPP SPECT and measurement of HOMA-IR as a parameter of insulin resistance.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2001-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Cardiac death

SECONDARY OUTCOMES:
All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Toshihiko Ono, MD, Study Director — Toujinkai Group
Locations (1):
- Toujinkai Hospital, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Nishimura M, Okamoto Y, Takatani T, Sato N, Nishida M, Hashimoto T, Yamazaki S, Kobayashi H, Ono T. Improvement of myocardial fatty acid metabolism by oral nicorandil in hemodialysis patients without coronary artery disease. J Nephrol. 2015 Apr;28(2):227-34. doi: 10.1007/s40620-014-0125-5. Epub 2014 Jul 29. PMID 25070153